CLINICAL TRIAL: NCT02614404
Title: Effect of Imatinib on Suppression of Malaria Parasites in Patients With Uncomplicated Plasmodium Falciparum Malaria
Acronym: MIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HuLow (Industry)
Collaborators: Purdue University (Other); University of Turin, Italy (Other); Università degli Studi di Sassari (Other); Hue University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HuLow-201605
Record Dates: First submitted 2015-11-16; First posted 2015-11-25 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Plasmodium falciparum; Uncomplicated malarial; imatinib mesylate; antimalarials
MeSH Terms: conditions — Malaria, Falciparum | interventions — Imatinib Mesylate; benzene-1,4-diphosphonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imatinib combination therapy (Experimental): Administration of imatinib (400 mg/day) plus dihydroartemisinin (40 mg/day) plus piperaquine (320 mg/day) to uncomplicated adult male malaria patients. Normal health parameters will be monitored continuously to evaluate safety and the decrease in peripheral blood parasitemia with time will be quantitated to assess efficacy.
  Interventions: Drug: Imatinib combination therapy
- dihydroartemisinin plus piperaquine (Active Comparator): Administration of dihydroartemisinin (40 mg/day) plus piperaquine (320 mg/day) to uncomplicated adult male malaria patients. Normal health parameters will be monitored continuously to evaluate safety and the decrease in peripheral blood parasitemia with time will be quantitated to assess efficacy.
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Imatinib combination therapy — Imatinib plus dihydroartemisinin plus piperaquine
  Other Names: Gleevec; Glivec
  Arms: Imatinib combination therapy
Drug: Dihydroartemisinin-piperaquine — Standard of care
  Other Names: Artekin; Eurartesim; Diphos; Timequin; Duocotecxin; Malacur; Ridmal
  Arms: dihydroartemisinin plus piperaquine

SUMMARY:
The purpose of this study is to determine the efficacy and safety of imatinib in combination with dihydroartemisinin plus piperaquine in the treatment uncomplicated P. falciparum malaria in adult male patients.

DETAILED DESCRIPTION:
An exploratory study to examine the efficacy and safety of imatinib mesylate in combination with dihydroartemisinin plus piperaquine on suppression of parasitemia in patients with uncomplicated Plasmodium falciparum malaria. In vitro studies of P. falciparum parasitized erythrocytes demonstrate that inhibitors of the protein tyrosine kinase SYK prevent malaria parasite egress from infected red blood cells and thereby terminate the parasite's life cycle. Although no potent syk kinase inhibitors were approved for human use at the time of initiation of this study, a bcr-abl tyrosine kinase inhibitor (imatinib mesylate (Gleevec®)) that also exhibits off-target inhibition of syk tyrosine kinase, has been FDA-approved for treatment of a number of human malignancies including chronic myelogenous leukemia and GIST. Because imatinib can be taken daily for many years without significant toxicity, it can be used to obtain a preliminary indication of whether inhibition of erythrocyte syk kinase can suppress parasitemia in patients with P. falciparum malaria. In a phase 1 clinical trial on the same patient population, anti-malaria activity was observed with imatinib, with little or no accompanying toxicity. Because dihydroartemisinin plus piperaquine constitute the currently used standard-of-care therapy for malaria in Southeast Asia, the above trial will test the safety and efficacy of the combination of imatinib plus dihydroartemisinin and piperaquine in treatment of uncomplicated malaria. In this pilot study, the rate of decrease in peripheral blood parasitemia in 30 adult male patients with uncomplicated malaria will be compared to the same rate of decrease in parasitemia in 30 adult male patients treated solely with dihydroartemisinin plus piperaquine.

ELIGIBILITY:
Inclusion Criteria:

* Gender: only adults are selected for the trial; note that female subjects cannot be women of child-bearing age.
* Age: 18-50 years.
* Target disease: Uncomplicated Plasmodium falciparum malaria

Exclusion Criteria:

* symptoms and signs of complicated malaria
* including continuous high fever of over 390C, psychiatric disorders, confusion, other neurological symptoms, symptoms and signs of functional impairment of the organs such as lungs, kidneys or cardiovascular system;
* symptoms and signs of liver damage or kidney damage
* symptoms and signs of another complicating infection such as pneumonia, dengue fever, and other bacterial infection.
* P. falciparum > 25.000 / mm3
* WBC <4000 and >10.000 /mm3

  * RBC < 3.5x106/mm3
  * Platelets < 40.000 /mm3
* Hemoglobin < 10 g/dL
* ALT more than 200% of the upper limit (56 units/L)
* AST more than 200% of the upper limit (40 units/L)
* Blood creatine more than 75% of the upper limit (men: 1.2 mg/dL, women 1 mgdL)
* Serum total protein < 6 g/L
* Glycemia < 50 mg/dL> 200 mg/dL
* Standard urine test Serious alterations
* Concomitant treatments

Antimalarial Drugs Anticoagulant therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Time to Parasite Clearance | From baseline to the time point when the blood parasite count is zero (up to a maximum of 5 days)
  Parasite clearance was determined by assessing the parasite count in blood, using thin film, thick film and qPCR analysis
28-day Cure Rate | Day 28
  28-day cure rate was defined as the percentage of participants with blood parasite count of zero after 28 days of treatment and no evidence of recurrent infection with the same parasite genotype after reduction of the asexual parasitemia. Follow up after treatment will only be performed in the case of complete clearance of parasites at D5 due to Imatinib treatment.

SECONDARY OUTCOMES:
Frequency of adverse events | Within 1 week of beginning treatment with imatinib
  Adverse events (AEs) are defined as events possibly related to the study drug as judged by physician that occur within 1 week of beginning treatment with imatinib.
  1. Incidence, severity, drug-relatedness, seriousness of adverse events
  2. Laboratory values (biochemistry and haematology)
  3. Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Huynh D Chien, MD, PhD, Principal Investigator — Hue University; Francesco M Turrini, MD, PhD, Principal Investigator — University of Turin, Italy; Philip S Low, PhD, Principal Investigator — Purdue University
Locations (1):
- A Tuc, Hương Hóa, Quang Tri, Vietnam